CLINICAL TRIAL: NCT03861897
Title: Efficacy of Non-instrumental Pleural Chest Physiotherapy (KRP-NI) in Initial Management of Infectious Pleural Effusion
Brief Title: Efficacy of Non-instrumental Pleural Chest Physiotherapy
Acronym: KINEPANCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHRD1815
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Infectious Pleural Effusion
Keywords: Non instrumental physiotherapy; Physiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention KRP-NI + KM (Experimental): Realization of Non instrumental pleural chest physiotherapy and Mobilization physiotherapy sessions (KRP-NI)
  Interventions: Other: KRP-NI + KM
- Control KM (Active Comparator): Realization of mobilization physiotherapy sessions (KM)
  Interventions: Other: KM

INTERVENTIONS:
Other: KRP-NI + KM — Non instrumental pleural chest physiotherapy (KRP-NI), 2 sessions a day on weekdays and 1 session a day on weekends and mobilization physiotherapy (KM), 1 session per day except weekend during the hospitalization. The combination of the two physiotherapy is KRP-NI + KM. Afterward, 3 sessions per week, renewable until M3 of non instrumental pleural respiratory physiotherapy. If necessary the doctor can prescribe sessions of mobilization physiotherapy
  Arms: Intervention KRP-NI + KM
Other: KM — Mobilization physiotherapy (1 session per day except weekend) during the hospitalization. Afterward, if necessary the doctor can prescribe sessions of mobilization physiotherapy(KM).
  Arms: Control KM

SUMMARY:
The main purpose of this study is to assess efficacy of non instrumental pleural chest physiotherapy on the recovery of respiratory function, at hospital discharge or 15 days after beginning the pleural chest physiotherapy, compared to physiotherapy with standard mobilization, in patients with infectious pleural effusion, who have received usual medical treatment.

DETAILED DESCRIPTION:
Pleural effusions are defined by an abnormal amount of fluid in the pleural space. Those complicating a pneumonia are commonly encountered in pneumology departments, and their number are increasing. If not quickly treated, complications often occur: pleural adhesions, pleural thickening which can lead to a restrictive lung disease, or even to surgery. The average length of stay in hospital of this patients is 15 days. The management of infectious pleural effusion consists of removing the fluid from the pleural space (pleural puncturing or drainage), with or without fibrinolytics, antibiotics, and chest physiotherapy. Chest physiotherapy is often prescribed, but its benefits are largely based on empirical evidence. In the absence of recommendations, chest physiotherapy is done in heterogeneous ways, in France and abroad.

Pleural chest physiotherapy combines postural respiratory exercises, increased ventilation with dynamics expirations, and early inspiratory exercises, resulting in mobilization of pleura and pleural fluid. The hypothesis is that pleural chest physiotherapy thus makes it possible to fight against pleural effusion stagnation, to help resorption of pleural fluid, to limit formation of pleural adhesions and fixed restrictive lung disease. This should improve the recovery of respiratory function, and allow a shorter hospital stay, an improvement of the quality of life, earlier resumption of activities, and a reduction in the risk of complications.

ELIGIBILITY:
Inclusion Criteria:

* ≥ eighteen years old
* to be hospitalized for an infectious pleural outpouring
* to have a liquid pleural outpouring diagnosed by echography or to scan thoracic
* presence of a Exudate according to the criteria of Light, to have at least criteria:

  * The ratio of pleural fluid protein to serum protein is greater than 0.5
  * The ratio of pleural fluid Lactate dehydrogenase (LDH) and serum LDH is greater than 0.6
  * The rate of pleural fluid LDH is > 2/3 upper limit of normal serum LDH of the laboratory concerned
* presence of at least two of the following criteria:

  * fever higher or equal 38°C (100.4°F)
  * thoracic pain
  * purulent sputum
  * purulent pleural effusion at the time of the exploring pleural puncture
  * hearth of crackling to the sounding
  * Inflammatory syndrome (CRP>15 mg/l and/or White blood cell >10 000 /mm3)
  * no known radiological hearth before
* Having undergone an evacuation gesture going back to less forty-eight hours: evacuation pleural puncture or repeated pleural punctures or pleural drainage allowing the evacuation of at least 100cc of pleural fluid
* Informed and having given its free, lit and express assent
* Patients with affiliation to the social security system

Exclusion Criteria:

* Patient having undergone a thoracotomy or thoracoscopy in the six previous months
* Patient having a pneumothorax
* Patient reached of a tuberculosis
* Patient unable to carry out a measurement of the vital capacity by portable spirometer at the inclusion
* Pregnant woman or nursing
* Patient having a life expectancy lower than three months
* Proven or suspected pleural neoplasia disease
* Patient hemodynamically unstable
* Patient having a respiratory insufficiency requiring the introduction of an artificial ventilation
* Patient carrying a chronic respiratory insufficiency under non-invasive ventilation with the long course
* Patient unable to carry out the exercises of physiotherapy (problem of communication and/or comprehension and/or physical inaptitude)
* Patient transplanted of a solid body, allograft or autograft of hematopoietic stem cells
* Patient with a seropositivity for the known HIV and cluster of differentiation 4 (CD4) <250/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Variation of vital capacity theoretical between the first day of inclusion and J15 or the last day of hospitalization | At 15 days after inclusion or the last day of hospitalization
  The Primary Outcome Measure is the variation of the percentage of vital capacity theoretical between the first day of inclusion and J15 or the last day of hospitalization using a portable spirometer (Spirobank II basic).
  Realized by an appraiser not being aware of the arm of randomization.

SECONDARY OUTCOMES:
Variation of vital capacity theoretical at M1,5 and M3 | At 3 months
  The variation of the percentage of vital capacity theoretical between the first day of inclusion and a month and half afterwards and between the first day of inclusion and three months afterwards using a portable spirometer (Spirobank II basic).
Measures the intensity of the pain: analogue visual scale | At 3 months
  Intensity of the pain with an analogue visual scale (AVS) at J15 or the last day of hospitalization, at one month and half after the first day of inclusion and at three months.
  The score is between 0 and 10. 0 is the best value (No pain) and 10 the worst (Maximum pain imaginable).
  Realized by an appraiser not being aware of the arm of randomization.
Measurement of rest dyspnea rated according to the modified Borg modified scale | At 3 months
  Measurement of the dyspnea of rest according to the scale of Borg modified at J15 or the last day of hospitalization, at one month and half after the first day of inclusion and at three months. The score is between 0 and 10. 0 is the best value (No shortness of breath) and 10 the worst (Maximum breathlessness).
  Realized by an appraiser not being aware of the arm of randomization.
Measurement of effort dyspnea rated according the mMRC scale | At 3 months
  Measurement of effort dyspnea rated according the Medical Research Council scale (mMRC) at J15 or the last day of hospitalization, at one month and half after the first day of inclusion and at three months.he score is between 0 and 4. 0 is the best value and 4 the worst.
  Realized by an appraiser not being aware of the arm of randomization.
Measure of quality of life: Respiratory Questionnaire St Georges | At one month and half
  Measure of quality of life with the Respiratory Questionnaire St Georges
Analysis of the thoracic scanner | At 3 months
  Centralized review of thoracic Scanner made at 3 months by radiologist who does not know the arm.
  Analysis of pleural pockets number and the maximum thickness of the pleural
Days of hospitalization | At 3 months
  Number of hospitalization days starting from inclusion
Proportions of complications at M3 | At 3 months
  Early proportions of complications, surgical treatment and death related to the infectious pleural outpouring.
Duration of sick leave | At 3 months
  Number of sick days accumulated in patients with a professional activity
Follow-up of physiotherapy carried out in the city | At 3 months
  For the intervention group : the number, the frequency and duration of the meetings of pleural chest physiotherapy carried out in a liberal physiotherapist and the use or not of an instrumental help
Opinion of the physiotherapist | At 3 months
  Measurement of the opinion and satisfaction of hospital and liberal physiotherapist participating by self-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique MONTRELAY, Principal Investigator — Hôpital NOVO
Locations (11):
- France (11):
  - Centre Hospitalier Universitaire Angers, Angers
  - Hôpital Victor Dupuy, Argenteuil
  - Hôpital de la Cavale Blanche, Brest
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier Intercommunal - Créteil, Créteil
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Groupe Hospitalier de la Rochelle, La Rochelle
  - Hôpital Dupuytren, Limoges
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Centre Hospitalier René Dubos, Pontoise

IPD SHARING:
Plan to Share IPD: No